CLINICAL TRIAL: NCT04765696
Title: Prospective RELOC-AGE: How Do Housing Choices and Relocation Matter for Active Ageing?
Acronym: RELOC-AGE
Status: Active, not recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); The Swedish Research Council (Other Government); Ribbingska Foundation in Lund (Unknown); Riksbyggen (Unknown); Karlshamnsbostäder AB (Unknown); Örebrobostäder (Unknown)
Responsible Party: Principal Investigator, Susanne Iwarsson, Professor, Lund University
Other Study IDs: 2020-03457
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Active Ageing
Keywords: Housing; Relocation; Health; Neighbourhood; Life space mobility; Housing preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons 55 years or older considering relocation: No intervention is administered.
  Interventions: Other: No intervention is administered

INTERVENTIONS:
Other: No intervention is administered — No intervention is administered, the cohort is followed in order to evaluate the impact of housing and relocation on active ageing outcomes.

SUMMARY:
The objective of prospective RELOC-AGE is to study housing choices and relocation and to examine the effects on active ageing among people aged 55+ considering relocation. All data collection will be conducted at baseline and after 1, 3, 5 and 7 years of follow-up.

DETAILED DESCRIPTION:
The objective of prospective RELOC-AGE is to study housing choices and relocation and to examine the effects on active ageing among people aged 55+ considering relocation.

Research Questions

1. What aspects of housing, health and participation predict a) relocation to different housing options in the ordinary housing stock; b) residential care facilities; c) remaining in the present dwelling?
2. How is the complex interaction between objective and perceived aspects of housing, health and participation associated with active ageing, and what are the patterns and characteristics of such dynamics?
3. What housing attributes do people aged 55+ considering relocation find important, and to what extent, when making their decisions on housing preferences?
4. How do people aged 55+ considering relocation reason a) regarding different housing options; b) motives for considering and effectuating relocation, and; c) to what extent are their motives fulfilled?

The sample will include people aged 55+ considering relocation. Recruitment will be made from a sub-sample based on waiting lists (n=22 000) among three housing companies in Sweden: Karlshamnsbostäder AB, Örebrobostäder AB, and Riksbyggen. The expected final sample size is n=3000. Quantitative data will be collected through a web survey and one telephone interview at baseline (2021) and by a web survey at follow-ups 2022, 2024, 2026 and 2028. Data on primary and secondary outcomes are based on established questionnaires used in previous research on older people, health, and housing as well as in national public health surveys in Sweden. In addition to primary and secondary outcomes (presented below), the surveys include demographic and socioeconomic characteristics including civil status, education level, economic situation, occupational status, holding a driver license, critical life events (e.g., death of spouse, long-term disease, divorce), original nationality; questions about present housing situation (dwelling characteristics (e.g., type and size of dwelling, location) and neighborhood characteristics (e.g., access to services and green areas), potential and realized mobility, social/cohabiting situation, time spent at home, housing adaptations); use of technical aids for mobility, use of health, social and informal care, thoughts about future housing, reasons related to consideration about relocating and moving intentions. Data on stated preferences in relation to housing will be collected in a specific survey based on a discrete choice methodology. Qualitative interviews will be conducted consecutively with a subsample (n=100) of respondents who have relocated during the follow-up period. Further, linking to register data will be made within the scope of Register RELOC-AGE, which is another part of the larger project.

For quantitative data, descriptive, exploratory, and inferential statistics will be used. For longitudinal analyses, generalized linear models or Cox regression with time-dependent covariates will be applied. Throughout, we will control for demographic and socioeconomic characteristics and other potential confounders and compare the results across different cohorts. Quantitative analyses will be conducted using standard statistical software. For analyses of DCE data, we will use the conditional logit model (also referred to as the multinomial logit model) as the reference model, but the analysis will be extended to mixed logit and latent class models to take preference heterogeneity into account. Qualitative interviews will be audio-recorded and transc¬ribed verbatim and principles from Grounded Theory will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Persons 55 years or older, living in Sweden, listed for relocation at any of the three housing companies Karlshamnsbostäder and Örebrobostäder (public housing companies) and Riksbyggen (a condominium provider)

Exclusion Criteria:

* Severe cognitive impairments or insufficient language skills to give informed consent and participate in telephone interviews

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons 55 years or older, living in Sweden, listed for relocation at any of the three housing companies Karlshamnsbostäder and Örebrobostäder (public housing companies) and Riksbyggen (a condominium provider)
Sampling Method: Probability Sample
Enrollment: 1964 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
University of Jyväskylä Active Aging Scale (UJACAS) | Change from Baseline Active Ageing score to 12 months
  17 items(areas of activity), each to be self-rated regarding goals, ability, autonomy and activity (total scores 0-272)
University of Jyväskylä Active Aging Scale (UJACAS) | Change from Baseline Active Ageing score to 36 months
  17 items(areas of activity), each to be self-rated regarding goals, ability, autonomy and activity (total scores 0-272)

SECONDARY OUTCOMES:
Life-space mobility | Change from Baseline Life-space mobility to 12 months
  6 items related to life spaces visited during the past four weeks, whether the person had visited (yes/no), frequency on a four-point scale, and level of dependence on others or technical equipment on a three-point scale)
Life-space mobility | Change from Baseline Life-space mobility to 36 months
  6 items related to life spaces visited during the past four weeks, whether the person had visited (yes/no), frequency on a four-point scale, and level of dependence on others or technical equipment on a three-point scale)
Meaning of home | Change from Baseline Meaning of home scores to 12 months
  28 items with statements to which respondents state agreement on a ten-point scale from 1 (not at all) to 10 (very much)
Meaning of home | Change from Baseline Meaning of home scores to 36 months
  28 items with statements to which respondents state agreement on a ten-point scale from 1 (not at all) to 10 (very much)
Housing related control beliefs | Change from Baseline Housing related control beliefs scores to 12 months
  24 items with statements to which respondents state agreement on a five-point scale from 1 (not at all) to 5 (very much)
Housing related control beliefs | Change from Baseline Housing related control beliefs scores to 36 months
  24 items with statements to which respondents state agreement on a five-point scale from 1 (not at all) to 5 (very much)
Usability in my home | Change from Baseline Usability in my home scores to 12 months
  4 items (selected from original instrument) with statements about aspects of usability rated on a five-point scale from 1 (not at all) to 5 (very much)
Usability in my home | Change from Baseline Usability in my home scores to 36 months
  4 items (selected from original instrument) with statements about aspects of usability rated on a five-point scale from 1 (not at all) to 5 (very much)
Housing satisfaction | Change from Baseline Housing satisfaction scores to 12 months
  One item "Are you happy with the condition of your home?" answered on a five-point scale from 1 (definitely not) to 5 ('yes, definitely)
Housing satisfaction | Change from Baseline Housing satisfaction scores to 36 months
  One item "Are you happy with the condition of your home?" answered on a five-point scale from 1 (definitely not) to 5 ('yes, definitely)
Health-related Quality of life | Change from Baseline Health-related Quality of Life to 12 months
  EuroQol-5d questionnaire (5 items, range 1-5 per item, with higher score indicating worse outcome)
Health-related Quality of life | Change from Baseline Health-related Quality of Life to 36 months
  EuroQol-5d questionnaire (5 items, range 1-5 per item, with higher score indicating worse outcome)
Self-rated health | Change from Baseline Self-rated Health to 12 months
  One item "How would you rate your own health", rated from 1 (bad) to 5 (excellent)
Self-rated health | Change from Baseline Self-rated Health to 36 months
  One item "How would you rate your own health", rated from 1 (bad) to 5 (excellent)
Life satisfaction | Change from Baseline Life satisfaction to 12 months
  One item "How satisfied are you with life in general", rated from 1 (very unsatisfied) to 6 (very satisfied)
Life satisfaction | Change from Baseline Life satisfaction to 36 months
  One item "How satisfied are you with life in general", rated from 1 (very unsatisfied) to 6 (very satisfied)
Housing enabler, functional limitations | Change from Baseline Functional limitations to 12 months
  8 items indicating presence (yes or yes to some extent) /absence (no) functional limitations
Housing enabler, functional limitations | Change from Baseline Functional limitations to 36 months
  8 items indicating presence (yes or yes to some extent) /absence (no) functional limitations
General self-efficacy | Change from Baseline Genreal Self-efficacy to 12 months
  10 items with statements to which respondents state agreement on a four-point scale from 1 (completely disagree) to 4 (totally agree)
General self-efficacy | Change from Baseline Genreal Self-efficacy to 36 months
  10 items with statements to which respondents state agreement on a four-point scale from 1 (completely disagree) to 4 (totally agree)
Physical exercise | Change from Baseline physical exercise duration/week to 12 months
  Rated as duration per week on five levels from 0 minutes to 2 hours or more
Physical exercise | Change from Baseline physical exercise duration/week to 36 months
  Rated as duration per week on five levels from 0 minutes to 2 hours or more
Physical activity | Change from Baseline physical activity duration/week to 12 months
  Rated as duration per week on six levels from 0 minutes to 2 hours or more
Physical activity | Change from Baseline physical activity duration/week to 36 months
  Rated as duration per week on six levels from 0 minutes to 2 hours or more
Frailty (FRESCH) | Change from Baseline Frailty scores to 12 months
  4 items to be answered yes or no
Frailty (FRESCH) | Change from Baseline Frailty scores to 36 months
  4 items to be answered yes or no
Satisfaction with mobility opportunities | Change from Baseline Satisfaction with mobility opportunities to 12 months
  One item, rated from 1 (very satisfied) to 5 (very unsatisfied)
Satisfaction with mobility opportunities | Change from Baseline Satisfaction with mobility opportunities to 36 months
  One item, rated from 1 (very satisfied) to 5 (very unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Malmgren Fänge, PhD, Study Chair — Lunds University
Locations (1):
- Active and Healthy Ageing Research Group, Department of Health Sciences Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zingmark M, Nordestrom F, Iwarsson S. Challenges related to self-assessment of active ageing during the Covid-19 pandemic in Sweden. BMC Res Notes. 2022 May 13;15(1):171. doi: 10.1186/s13104-022-06059-3. PMID 35562784
- [Derived] Zingmark M, Bjork J, Granbom M, Gefenaite G, Nordestrom F, Schmidt SM, Rantanen T, Slaug B, Iwarsson S. Exploring Associations of Housing, Relocation, and Active and Healthy Aging in Sweden: Protocol for a Prospective Longitudinal Mixed Methods Study. JMIR Res Protoc. 2021 Sep 21;10(9):e31137. doi: 10.2196/31137. PMID 34546172
- See also: Project website — https://www.case.lu.se/forskning/relocage